CLINICAL TRIAL: NCT06531239
Title: Relationship of Motor Competence, BMI and Physical Fitness of School Going Children
Brief Title: The Link Between Motor Competence BMI and Physical Fitness School-age Children
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR&AHS/23/0783
Record Dates: First submitted 2024-06-11; First posted 2024-07-31 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Children, Only
Keywords: Physical fitness.; BMI; Motor competence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The term "physical fitness" in youngsters describes their general health and capacity for movement. It consists of elements including flexibility, muscular strength and endurance, cardiovascular endurance, and body composition. Children that are physically fit can run, jump, climb, and play without becoming fatigued easily. The body mass index is a metric used to determine how much a person weighs in connection to their height.

Motor competence assesses an individual's ability to accomplish various motor skills and movements. The project aims to study the development and competency of motor skills, as well as factors influencing them, such as physical fitness and training. A cross sectional study will be conducted in different schools of Lahore through convenient sampling. Data will be gathered from a healthy population of age 5 to 8 years. Children with dementia and other mental disorders are excluded. BMI and IPAC-SF tools are used for data collection. Various types of physical activities including walking, moderate intensity and vigorous intensity exercises are used. Data will be analyzed by SPSS 26 version.

DETAILED DESCRIPTION:
The healthy outcomes of a group of individuals, including the distribution of such outcomes within the group," and we argue that the field of population health includes health outcomes, patterns of health determinants, and policies and intervention .Motor competence (MC) is defined as proficiency in fundamental motor skills including locomotor and object control skills, and represents the degree of skilled performance in a wide range of motor tasks as well as the movement quality, coordination and control underlying a particular motor outcome. Engagement in physical activity in the early years of childhood is associated with lower adiposity levels, higher cognitive performance besides improved psychosocial and cardiometabolic health. Many schools in Pakistan mainly concentrates on the higher study level and very low attention towards children's physical health that may impair due to low physical activity level and increased sedentary behavior leading to obesity and other health issues. Recently, increased interest has been shown by the researcher and investigators in the prevalence of adiposity, inactivity, and health risk factors among adolescents, and the appearance of cardiovascular, neuromuscular, and metabolic diseases during adolescence emphasized the necessity to consider physical activity and physical fittness vital in the growth of adolescent children. physical fitness refers to the ability of your body systems to work together efficiently to allow you to be healthy and perform activities of daily living . Health-related components of Physical Fitness. There are five components of physical fitness: . body composition, flexibility, muscular strength, muscular endurance, and cardiorespiratory endurance. Stodden et al. put forth a conceptual model describing the dynamics between physical activity and other healthrelated factors that lead to a positive spiral of engagement or a negative spiral of disengagement in physical activity. The outcomes of a BMI test might be classified as underweight, normal weight, overweight, or obese common interpretation is that it represents an index of an individual's fatness. In addition, it is widely used in determining public health policies. It is calculated by dividing the person's weght in kilogram by the square of their height in meters. Physical fitness was measured using the International Physical Activity Questionnaire-Short Form (IPAQ-SF), which contains seven questions. The questionnaire was used to obtain the total minutes of physical activity per week and sitting time per day. PMC tool assesses the performance of six locomotors and seven object control skills with a total raw score of 100. Three locomotion tasks (i.e., running, skipping ,and jumping) and three ball skill tasks (i.e., catching, overhand throw, and underhand throw) were selected to represent locomotion and object control capacities, respectively. Before the assessment of each skill, a trained researcher first demonstrated the skill, and the participants were allowed one practice trial. BMI (Body mass index) is a common method used to measure obesity. Waist circumference, neck circumference, waist-to-hip ratio, skinfold thicknesses.

ELIGIBILITY:
Inclusion Criteria:Children between the ages of 5 and 8 years .

* Male and female will be included.
* BMI citatory normal, overweight, underweight, obese.

Exclusion Criteria:

* Children with Diabetes

  * Children with any physical or cognitive disabilities that would significantly impact motor competence.
  * abnormal visual and neurological development .
  * BMI citatory normal, overweight, underweight, obese excluded.
  * cardiovascular and respiratory chronic diseases.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Data will be measured through BMI, motor competence and physical activity under the sample size 271 and age of children 5 to 8 years
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 8 weeks
  To calculate BMI weight machine will be used height we use inches tap in inches and converted it into meters respectively.
Physical fitness | 8 weeks
  International Physical Activity will be used Questionnaire - Short Form. The questionnaire asks about the frequency and time of various types of physical activities, including walking, moderate-intensity activities, and vigorous-intensity activities. There are two forms of output from scoring the IPAQ.mild one, moderate two, severe three.
Motor competence | 8 weeks
  locomotion skills (run, gallop, hop, leap, horizontal jump, slide), and six object control will be used

CONTACTS AND LOCATIONS:
Overall Officials: Rimsha Majid, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silberberg M, Martinez-Bianchi V, Lyn MJ. What Is Population Health? Prim Care. 2019 Dec;46(4):475-484. doi: 10.1016/j.pop.2019.07.001. Epub 2019 Jul 31. PMID 31655744